CLINICAL TRIAL: NCT06129045
Title: Effects of Sleep Hygiene Education on Sleep Health in Adults Ages 50-80
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Ashley Pfeiffer, Associate Professor, Black Hills State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHSU; P20GM103443 (NIH)
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Sleep Hygiene
Keywords: Behavior Change; Older adults; sleep hygiene
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Three arm study: No intervention, video only, video plus text messaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group One, Video (Experimental): One-time sleep hygiene education
  Interventions: Behavioral: One-time educational video
- Group Two, Video Plus Texts (Experimental): One-time sleep hygiene education plus repeated education through automated text messaging
  Interventions: Behavioral: Educational video plus repeated education
- Group Three, (No Intervention): Control group with no intervention assigned

INTERVENTIONS:
Behavioral: One-time educational video — Sleep hygiene educational tips provided through a video participants watch on their own.
  Arms: Group One, Video
Behavioral: Educational video plus repeated education — Sleep hygiene educational tips are provided first through a video participants watch on their own and then tips are repeated through daily automated text messaging for an additional 4 weeks.
  Arms: Group Two, Video Plus Texts

SUMMARY:
This will be a study looking at trying to change older adults' behavior in regard to good sleep hygiene practices. Investigators will assess the efficacy through subjective outcome measures and objective physiological markers of good sleep through data collected with wearable technology devices.

DETAILED DESCRIPTION:
Older adults ages 50-80 will be recruited and placed into one of three groups. Group One will watch a one-time educational video on sleep hygiene, Group Two will watch the video plus be sent daily automated text messages to reinforce the education learned in the video, and Group Three will be a control group with no intervention. The participants in Groups One and Two will receive the education after two weeks of data tracking on a Fitbit device. They then will have four additional weeks of tracking. At the end of the study time of six weeks, all participants will return for follow-up testing. The sleep tracker will monitor the physiological markers of sleep provided by wearable technology on sleep efficiency, time in bed, time actually sleeping, and time spent at each stage of sleep.

ELIGIBILITY:
Inclusion Criteria:

* own a smartphone with the capability of receiving text messages.

Exclusion Criteria:

* an untreated diagnosed sleep disorder such as insomnia or obstructive sleep apnea
* inability to wear the device on their wrist

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Pfeiffer, DPT, Principal Investigator — Black Hills State University
Locations (1):
- Black Hills State University, Spearfish, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We recruited 125 participants who completed the informed consent and intial evaluation. Six participants dropped out due to personal reasons leaving 119 participants that were able to see the study through to the conclusion. Funding ran out prior to being able to recruit any additional participants.
Period: Overall Study
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Started | 40 | 42 | 43
Completed | 39 | 41 | 39
Not Completed | 1 | 1 | 4
Not completed — Lost to Follow-up | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three, | Total
Number analyzed (Participants) | 39 | 41 | 39 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.2) | 66.7 (6.1) | 66.3 (7.4) | 66.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 31 | 24 | 78
  Male | 16 | 10 | 15 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 36 | 40 | 39 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 41 | 39 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0
Readiness to change sleep behavior 0-10 visual analog scale [Mean (Standard Deviation); unit: units on a scale] — Each participant was asked, "How ready are you to change your sleep behaviors?" They were given a scale from 0, which read "not at all ready to change sleep behaviors" and then had options of 1,2,3,4,5,6,7,8,9, and 10. 10 read "completely ready to change sleep behaviors." Each participant chose which number most reflected where they were at on their readiness to change their sleep behaviors at that current moment in time. 0 indicated they weren't feeling ready, and 10 indicated feeling completely ready. Population: The average score on the readiness to change 0-10 scale is documented below for each intervention group.
  units on a scale | 5.97 (3.30) | 7.02 (3.00) | 6.43 (2.89) | 6.49 (3.07)

OUTCOME MEASURES:

1. Primary Outcome: Change Score of Pittsburgh Sleep Quality Index
Description: Change Score From Baseline to 6-week Follow up on the Pittsburgh Sleep Quality Index. Outcome measure for quality of sleep. Score ranges 0-21 with higher score equaling poor sleep quality
Time Frame: 6-weeks
Population: One person did not complete the PSQI on follow-up in the video only group due to technology error.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 38 | 41 | 39
Score on a scale | 1 (3.01) | 1.12 (2.87) | -0.615 (3.02)

2. Primary Outcome: Change Score of Sleep Hygiene Index
Description: Change Score From Baseline to 6-week Follow up on the Sleep Hygiene Index. Outcome measure for good sleep hygiene. Scores range from 0-52. Higher scores equate to worse sleep hygiene.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 39 | 41 | 39
score on a scale | 2.41 (5.79) | 1.97 (5.29) | .64 (3.78)

3. Primary Outcome: Change Score of Epworth Sleepiness Scale
Description: Change Score From Baseline to 6-week Follow up on the Epworth Sleepiness Scale. Outcome measure for daytime sleepiness. Score ranges 0-24 with higher score equaling worst daytime sleepiness.
Time Frame: 6 week period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 39 | 41 | 39
score on a scale | 1.6 (3.3) | 1.71 (2.1) | 0.39 (3.5)

4. Primary Outcome: Change Score Total Sleep Time
Description: The average total sleep time per night in minutes for each participant was recorded.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 39 | 41 | 39
minutes per night | -2.9 (52.9) | 8.24 (56.9) | -4.3 (45.4)

5. Primary Outcome: Change Score for Total Time Awake
Description: The average total time awake per night in minutes for each participant was recorded.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 39 | 41 | 39
minutes per night | -2.9 (22.8) | -1.7 (12.7) | 2.3 (13.2)

6. Secondary Outcome: Change on the Perceived Stress Scale
Description: Outcome measure for average stress levels. Scores range from 0-40. The higher the score the worse the stress levels.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
Number analyzed (Participants) | 39 | 41 | 39
score on a scale | -0.11 (3.85) | 1.71 (4.51) | 0.23 (3.17)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, 6 week time period
Arm/Group | Group One, Video | Group Two, Video Plus Texts | Group Three,
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/39

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT06129045/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT06129045/SAP_001.pdf